CLINICAL TRIAL: NCT04890171
Title: Comparison of Endoscopic Resection and Surgery for Early Gastric Cancer With Undifferentiated Histological Type: a Multicenter Randomized Controlled Trial (ERASE-GC Trial)
Brief Title: Comparison of Endoscopic Resection and Surgery for Early Gastric Cancer With Undifferentiated Histological Type
Acronym: ERASE-GC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul St. Mary's Hospital, The Catholic University (Unknown); Chilgok Kyungpook National University Hospital (Unknown); Pusan National University Hospital (Other); Samsung Medical Center, Sungkyunkwan University School of Medicine (Unknown); Severance Hospital, Yonsei University College of Medicine (Unknown); Gangnam Severance Hospital, Yonsei University College of Medicine (Unknown); Asan Medical Center (Other); Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Il Ju Choi, Principal Scientist, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2021-0117
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stomach Cancer; Undifferentiated Type; Expanded Indication of Endoscopic Resection
Keywords: Early gastric cancer; Endoscopic submucosal dissection; Surgery; Undifferentiated type; Expanded indication
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic treatment arm (Active Comparator): Endoscopic submucosal dissection
  Interventions: Procedure: Endoscopic submucosal dissection
- Surgical treatment group (Active Comparator): Gastrectomy with lymph node dissection
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — Endoscopic submucosal dissection by a endoscopist using endoscopic devices
  Arms: Endoscopic treatment arm
Procedure: Surgery — Gastrectomy with lymph node dissection by a surgeon
  Arms: Surgical treatment group

SUMMARY:
This multi-center, randomized controlled trial is designed to evaluate clinical effectiveness and cost-effectiveness of ESD for undifferentiated type of EGC meeting the expanded indication compared with surgery.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a minimally invasive treatment of early gastric cancer (EGC). Because of the stomach preservation, ESD provides a better quality of life (QoL) in EGC patients than surgery. In addition, medical costs are lower in patients underwent ESD than in those underwent surgery. In 2018, gastric cancer management guidelines by the Korean Gastric Cancer Association and Japanese Gastric Cancer Association (JGCA) stated that undifferentiated type of EGC, clinically diagnosed as tumor confined to the mucosa without ulcer, and size ≤2 cm, is included in the expanded indication of ESD. In the 2018 JGCA guideline (version 5), ESD is an investigational treatment for patients with undifferentiated type of EGC meeting the expanded indication whereas surgery (gastrectomy with lymph node dissection) is a standard treatment. Previous single center retrospective studies reported favorable long-term outcomes of ESD for undifferentiated type EGC meeting the expanded criteria on final pathological evaluations compared with that of surgery. More recently, a multi-center retrospective cohort study including 18 Korean university hospitals also reported no significant difference in overall mortality between ESD and surgery after propensity score matching (hazard ratio [HR] for overall mortality in the ESD group, 2.36; 95% confidence interval [CI] 0.91-6.10; p=0.078) during a median follow-up of 75.6 months. However, gastric cancer recurrence occurred only in the ESD group, and the HR for gastric cancer recurrence in the ESD group was 25.49 (95% CI 1.32-491.27; p=0.032). The 3-year disease-free survival (DFS) rate including gastric cancer recurrence or death was 94.9% in the ESD group and 98.1% in the surgery group. Thus, surgery group had a better DFS than ESD group (p=0.002 by log-rank test), and the HR for gastric cancer recurrence or death in the surgery group compared with the ESD group was 0.26 (95% CI, 0.10-0.64; p=0.003). However, previous studies could provide only a low level of evidence because of study limitations including the retrospective study design and incomplete data of patient survival and gastric cancer recurrence during follow-up. The studies did not evaluate QoL and cost-effectiveness after ESD and surgery. Therefore, we designed a multi-center, randomized controlled trial to provide a high level of evidence for clinical effectiveness and cost-effectiveness of ESD for undifferentiated type of EGC meeting the expanded indication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with undifferentiated type EGC (signet ring cell carcinoma, poorly differentiated tubular adenocarcinoma, or poorly cohesive carcinoma) that meets the expanded indication of ESD 1) Tumor confined to the mucosa without ulcer, and size ≤2 cm on endoscopic evaluations 2) No evidence of lymph node metastasis and distant metastasis on abdominal CT scan
2. Adult patients aged 19-75 years
3. Patients who had willingness to sign an informed consent form

Exclusion Criteria:

1. Patient age: < 19 years or age > 75 years
2. Diagnosis and active treatment for other organ cancer except carcinoma in situ and non-melanomatous skin cancer within 5 years
3. Previous gastrectomy or esophagectomy history
4. Multiple gastric cancers
5. Current treatment for serious medical condition which could hinder study participation including severe heart dysfunction, liver cirrhosis, renal failure, chronic obstructive pulmonary disease or asthma, or uncontrolled infection
6. Inability to provide an informed consent
7. Inadequate conditions for study enrollment according to the evaluation of study physicians

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival in the ITT population | 3 years after the last participant enrollment
  Disease-free survival (gastric cancer recurrence or death from any causes)

SECONDARY OUTCOMES:
3-year disease-free survival in the PP population | 3 years after the last participant enrollment
  Disease-free survival (gastric cancer recurrence or death from any causes)
Overall survival | 5 years after the last participant enrollment
  Overall survival (death from any causes)
Curative resection rate of ESD | 2 year after the participant enrollment
  Curative resection on the final pathological evaluation
Quality of life changes during follow-up periods | 3 years after the last participant enrollment
  QoL changes using questionnaire
Treatment related complications (adverse events) | 3 years after the last participant enrollment
  Early (within 30 postoperative days) and late complications (after 30 postoperative days)
Cost-effectiveness measured with Incremental cost effective ratio (ICER) | 3 years after the last participant enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea